CLINICAL TRIAL: NCT03784820
Title: Targeting Relationship Domains in Community-Based Treatment of Binge-Eating Disorder
Brief Title: Uniting Couples in the Treatment of Binge-Eating Disorder
Acronym: UNITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-1379; 1R34MH113681-01A1 (NIH)
Record Dates: First submitted 2018-12-19; First posted 2018-12-24 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-03

CONDITIONS: Binge-Eating Disorder
Keywords: Binge-Eating Disorder; Eating disorders; Couple therapy; CBT
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either couple therapy (UNITE) or individual therapy (CBT-E) for binge-eating disorder and will receive 16 1-hour sessions of the respective treatment. All study hypotheses will be tested using recommended Intent-To-Treat (ITT) methods. Differential treatment effects in individual functioning variables will be tested using 2 (time) x 2 (treatment) mixed-effect ANOVAs for binge-purge frequency and eating disorder outcomes and 2 (partner) x 3 (time) x 2 (treatment) mixed-effect ANOVAs for psychological outcomes. (Some variables will have 4 time points). Differential treatment effects in target relationship variables will be tested using 2 (partner) x 2 (time) x 2 (treatment) mixed-effect ANOVAs for all outcomes except vocally encoded emotional arousal. Differential treatment effects of vocally encoded emotional arousal will be tested using repeated-measures Actor Partner Interdependence Models (RM-APIMS).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UNITE (Experimental): UNITE is a manualized cognitive-behavioral couple therapy (CBCT) intervention that engages the couple to address the core psychopathology of BED.
  Interventions: Behavioral: UNITE
- CBT-E (Active Comparator): CBT-E is a trans-diagnostic cognitive behavioral individual therapy treatment for eating disorders. It has been shown to be effective in numerous controlled and open trials.
  Interventions: Behavioral: CBT-E

INTERVENTIONS:
Behavioral: UNITE — UNITE includes three stages: early treatment (psychoeducation and understanding the couple's experience of BED within the relationship); mid-treatment (effective communication, interpersonal problem-solving, and emotion regulation skills), and late treatment (relapse prevention). Additional relevant topics may be covered including body image, weight stigma, weight and health concerns, and intimacy and sexuality issues.
  Arms: UNITE
Behavioral: CBT-E — CBT-E includes four stages: an introductory stage (psychoeducation, normalization of eating patterns, and symptom self-monitoring); a second, brief stage (review progress and formulate plans for the subsequent treatment phase); a third stage (elimination of dieting, reducing shape checking and avoidance behaviors, educating about mood tolerance, and targeting overevaluation of shape and weight); and the fourth stage (maintaining progress and minimizing relapse risk).
  Arms: CBT-E

SUMMARY:
The purpose of this study is to test the feasibility, acceptability, and preliminary effectiveness of a novel couple-based intervention for binge-eating disorder (BED) relative to an established evidence-based individual treatment (cognitive-behavioral therapy-enhanced; CBT-E) in a community clinic setting.

DETAILED DESCRIPTION:
Clinicians' options for BED treatment are inadequate. Treatments for BED have demonstrated efficacy in controlled settings with specialist therapists and expert supervision, but much less in known about the effectiveness of BED interventions and whether the transition of evidence-based treatments to the community results in poorer outcomes. UNITE activates a key resource by incorporating an important part of the patient's social environment (the partner) into treatment. The investigators hypothesize that UNITE will show preliminary evidence of being superior to CBT-E in achieving binge abstinence via engaging ED-related relationship targets, including improved (a) communication around the disorder, (b) disorder-specific interpersonal problem-solving/ behavioral change skills, and (c) partner-assisted emotion regulation. The investigators will assess targeted relationship domains with observational and speech prosody measures during clinic interactions and self-reports reflecting experiences outside the clinic. Because the couple is learning how to work together to address BED, the investigators hypothesize that maintenance of gains will show evidence consistent with superiority in UNITE.

ELIGIBILITY:
Inclusion Criteria:

* current Diagnostic and Statistic Manual (DSM-5) criteria for binge-eating disorder (patient only)
* at least 18 years of age
* English speaking and able to read
* in a committed relationship for at least 6 months regardless of sexual orientation
* live with partner (or are interact with each other daily)
* partner willingness to participate in treatment
* able to travel to Chapel Hill, North Carolina weekly for treatment

Exclusion Criteria:

* alcohol or drug dependence in the past year
* current anorexia nervosa
* current significant suicidal ideation with active suicidal intent
* severe depression that would seriously interfere with functional capacity
* developmental disability that would impair the ability to benefit from the intervention
* any psychosis, schizophrenia, or bipolar I disorder, unless stably remitted on maintenance therapy for at least 1 year
* moderate to high reported levels of physical violence from either partner
* unwillingness to forgo non-protocol concurrent couple therapy or individual therapy (patient only)
* previously participated in the UNITE pilot trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Bulik, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Donald Baucom, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
It is our intention to make data available to the general scientific community at the conclusion of the clinical trial. Given the fact that most of the entities involved in this application must be HIPAA compliant, deidentification of data along HIPAA guidelines will guide the development of the final database to be shared. The current plan would be to have the dataset available via the web through postings of the information on the Academy for Eating Disorders, the Eating Disorders Research Society, and the Association for Behavioral and Cognitive Therapy websites. Data will be provided in SAS and SPSS formats. The investigators will provide a detailed protocol and a code book. The availability of the de-identified data on these web pages would be announced in journals and publications of interest to clinicians and researchers in the areas of eating disorders, couple therapy, and cognitive-behavioral therapy.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data as described above will be made available 12 months after publication of the primary outcome paper.
Access Criteria: IRB approval for secondary data analysis, an executed data sharing agreement with UNC-CH and approval by principal investigators.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between September 2018 to January 2021 from local physician offices, social media, advertisements, and local listservs. Potential participants were asked to contact the Research Coordinator for more information. Potential participants completed a screening questionnaire by phone with the Research Coordinator. The setting for the study was an outpatient clinic at the University of North Carolina at Chapel Hill.
Pre-assignment Details: After consenting to participate and completing an initial phone screening, participants were asked to complete a pre-treatment assessment consisting of electronic questionnaires and an in-person interview to determine study eligibility. The patient with binge-eating disorder (BED) in each couple had to provide written certification from their primary care provider (PCP) that their health status was suitable for this study. After determining eligibility, patients were randomized.
Groups:
- CBT-E - Patients; CBT-E - Partners: CBT-E is a trans-diagnostic cognitive behavioral individual therapy treatment for eating disorders. It has been shown to be effective in numerous controlled and open trials.
  CBT-E: CBT-E includes four stages: an introductory stage (psychoeducation, normalization of eating patterns, and symptom self-monitoring); a second, brief stage (review progress and formulate plans for the subsequent treatment phase); a third stage (elimination of dieting, reducing shape checking and avoidance behaviors, educating about mood tolerance, and targeting overevaluation of shape and weight); and the fourth stage (maintaining progress and minimizing relapse risk).
- UNITE - Patients; UNITE - Partners: UNITE is a manualized cognitive-behavioral couple therapy (CBCT) intervention that engages the couple to address the core psychopathology of BED.
  UNITE: UNITE includes three stages: early treatment (psychoeducation and understanding the couple's experience of BED within the relationship); mid-treatment (effective communication, interpersonal problem-solving, and emotion regulation skills), and late treatment (relapse prevention). Additional relevant topics may be covered including body image, weight stigma, weight and health concerns, and intimacy and sexuality issues.
Period: Overall Study
Arm/Group | CBT-E - Patients | CBT-E - Partners | UNITE - Patients | UNITE - Partners
Started | 11 | 11 | 11 | 11
Pre (T0) Intent-to-Treat (ITT) | 11 | 11 | 11 | 11
Mid-Treatment (T1) Intent-to-Treat (ITT) | 10 | 7 | 9 | 9
Post (T2) Intent-to-Treat (ITT) | 7 | 6 | 9 | 9
3 Month Fup (T3) Intent-to-Treat (ITT) | 6 | 6 | 9 | 9
6 Month Fup (T4) Intent-to-Treat (ITT) | 6 | 6 | 8 | 8
Pre (T0) Modified Intent-to-Treat (mITT) | 11 | 11 | 10 | 10
Mid-Treatment (T1) Modified Intent-to-Treat (mITT) | 10 | 7 | 8 | 8
Post (T2) Modified Intent-to-Treat (mITT) | 7 | 6 | 8 | 8
3 Month Fup (T3) Modified Intent-to-Treat (mITT) | 6 | 6 | 8 | 8
6 Month Fup (T4) Modified Intent-to-Treat (mITT) | 6 | 6 | 7 | 7
Completed | 6 | 6 | 8 | 8
Not Completed | 5 | 5 | 3 | 3
Not completed — Lost to Follow-up | 5 | 5 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Patients with binge-eating disorder and their partners who satisfied study inclusion and exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-E | UNITE | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.00 (11.97) | 40.27 (10.31) | 41.14 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Subtotals for patients and partners are provided.
  Participants
    Patients: number analyzed (Participants) | 11 | 11 | 22
    Patients: Female | 3 | 2 | 5
    Patients: Male | 8 | 9 | 17
    Partners: number analyzed (Participants) | 11 | 11 | 22
    Partners: Female | 7 | 8 | 15
    Partners: Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall number of participants is equal to the number of patients and partners combined.
  Participants
    Patients: number analyzed (Participants) | 11 | 11 | 22
    Patients: Hispanic or Latino | 1 | 1 | 2
    Patients: Not Hispanic or Latino | 10 | 10 | 20
    Patients: Unknown or Not Reported | 0 | 0 | 0
    Partners: number analyzed (Participants) | 11 | 11 | 22
    Partners: Hispanic or Latino | 0 | 1 | 1
    Partners: Not Hispanic or Latino | 11 | 10 | 21
    Partners: Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The overall number of participants is equal to the number of patients and partners combined.
  Participants
    Patients: number analyzed (Participants) | 11 | 11 | 22
    Patients: Race: White | 10 | 10 | 20
    Patients: Race: Other | 1 | 1 | 2
    Partners: number analyzed (Participants) | 11 | 11 | 22
    Partners: Race: White | 10 | 9 | 19
    Partners: Race: Other | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Modified Intent-to-Treat Patients With Binge-eating Abstinence
Description: Binge-eating abstinence is measured using the Eating Disorder Examination-Questionnaire (EDE-Q) and is the number of participants across study time points achieving abstinence from objective binge eating over the past 28 days. The EDE-Q measure replaces the measure in the protocol to capture a month of abstinence. The weekly binge measure was unsuitable upon review of the data because the 4 times weekly measures did not capture an exact 4-week time frame because of therapy scheduling irregularities, as verified by date-stamps of measure completion. Also, the weekly binge measure captured the past 7 days and was administered every session and once at other timepoints.
Time Frame: Mid-Treatment (after 8 weekly treatment sessions) (T1), Post (after 16 weekly treatment sessions) (T2), 3 Month Fup (T3), 6 Month Fup (T4)
Population: Only patients completed this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 10 | 8
Participants
  Mid-Treatment (T1) | 2 | 1
  Post (T2): number analyzed (Participants) | 7 | 8
  Post (T2) | 5 | 4
  3 Month Fup (T3): number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) | 5 | 5
  6 Month Fup (T4): number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) | 4 | 6
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.36, Mixed Models Analysis — Comparison of Patients at Post (T2) [CBT-E is the reference]; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.04 to 3.27]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.38, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3) [CBT-E is the reference]; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.02 to 4.60]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.54, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4) [CBT-E is the reference]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.18 to 27.39]

2. Secondary Outcome: Mean Binge-eating Frequency in Modified Intent-to-Treat Patients
Description: Binge-eating frequency is measured using the Eating Disorder Examination-Questionnaire (EDE-Q) number of objective binge episodes item which spans the past 28 days. Range is 0-no upper limit, with higher frequency indicative of more severe pathology. The EDE-Q measure replaces the originally planned measure in the protocol.
Time Frame: Pre (T0), Mid-Treatment (after 8 weekly treatment sessions) (T1), Post (after 16 weekly treatment sessions) (T2), 3 Month Fup (T3), 6 Month Fup (T4)
Population: Only patients completed this measure.
Measure: Mean (Standard Deviation); unit: number of binge-eating episodes
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 11 | 10
number of binge-eating episodes
  Pre (T0) | 12.45 (9.18) | 14.50 (15.30)
  Mid-Treatment (T1): number analyzed (Participants) | 10 | 8
  Mid-Treatment (T1) | 6.70 (5.31) | 3.88 (2.42)
  Post (T2): number analyzed (Participants) | 7 | 8
  Post (T2) | 1.00 (1.73) | 1.50 (1.85)
  3 Month Fup (T3): number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) | 0.83 (2.04) | 0.75 (1.16)
  6 Month Fup (T4): number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) | 0.50 (0.84) | 0.57 (1.51)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.52, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = 0.51, 95% CI 2-sided [-1.06 to 2.09]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.97, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = 0.04, 95% CI 2-sided [-1.99 to 2.07]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.59, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 0.62, 95% CI 2-sided [-1.66 to 2.89]

3. Secondary Outcome: Mean Eating Disorder Examination-Questionnaire (EDE-Q) Global Score in Modified Intent-to-Treat Patients
Description: Eating disorder symptomatology is measured using the Eating Disorder Examination-Questionnaire (EDE-Q) global score. This self-report questionnaire assesses the presence and degree of specific psychopathology associated with eating disorders over the previous 28 days. The global score is obtained by summing the four subscale scores (Restraint, Eating Concern, Shape Concern, and Weight Concern) and then dividing this sum by the number of subscales (i.e., four). The global score range is 0 - 6. Higher scores are indicative of greater eating disorder symptomatology (i.e., worse outcome).
Time Frame: as for outcome 2
Population: Only patients completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 11 | 10
score on a scale
  Pre (T0) | 2.97 (1.14) | 3.53 (0.68)
  Mid-Treatment (T1): number analyzed (Participants) | 10 | 8
  Mid-Treatment (T1) | 1.89 (1.16) | 2.81 (0.70)
  Post (T2): number analyzed (Participants) | 7 | 8
  Post (T2) | 1.77 (0.47) | 1.82 (0.63)
  3 Month Fup (T3): number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) | 1.38 (0.82) | 1.66 (0.79)
  6 Month Fup (T4): number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) | 1.18 (0.73) | 1.40 (0.45)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.86, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = 0.05, 95% CI 2-sided [-0.45 to 0.54]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.44, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = 0.30, 95% CI 2-sided [-0.46 to 1.06]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.36, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 0.31, 95% CI 2-sided [-0.36 to 0.98]

4. Secondary Outcome: Mean Binge-Eating Scale (BES) Total Score in Modified Intent-to-Treat Patients
Description: The Binge-Eating Scale is a 16-item self-report scale that assesses behavioral, affective, and attitudinal components of the subject experience of binge-eating. Item responses range from 0 to 3, with a total score range of 0 to 48. Higher sum scores indicate greater binge-eating severity and associated emotional distress.
Time Frame: as for outcome 2
Population: Only patients completed this measure. Participants who provided data were analyzed. Some participants provided partial data at study time points, explaining discrepancy(ies) between the mITT Participant Flow N and N analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 11 | 10
score on a scale
  Pre (T0) | 25.40 (6.60) | 28.83 (7.02)
  Mid-Treatment (T1): number analyzed (Participants) | 10 | 8
  Mid-Treatment (T1) | 15.17 (8.37) | 17.76 (6.20)
  Post (T2): number analyzed (Participants) | 7 | 7
  Post (T2) | 9.56 (4.60) | 11.30 (5.98)
  3 Month Fup (T3): number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) | 7.17 (6.37) | 8.17 (4.70)
  6 Month Fup (T4): number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) | 7.00 (8.10) | 9.64 (3.96)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.33, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = 2.47, 95% CI 2-sided [-2.54 to 7.49]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.46, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = 2.18, 95% CI 2-sided [-3.59 to 7.95]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.27, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 3.83, 95% CI 2-sided [-2.94 to 10.60]

5. Secondary Outcome: Mean Yale-Brown Obsessive-Compulsive Scale Modified for Binge-Eating (YBOCS-BE) Total Score in Modified Intent-to-Treat Patients
Description: The Yale-Brown Obsessive-Compulsive Scale Modified for Binge-Eating measures the obsession of binge-eating thoughts and compulsiveness of binge-eating behaviors. The scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms). The total score range is 0 to 40. Higher scores indicate greater severity of compulsive behaviors and preoccupations related to binge-eating.
Time Frame: Pre (T0), Mid-Treatment (after 8 weekly treatment sessions) (T1), Post (after 16 weekly treatment sessions) (T2), 6 Month Fup (T4)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 11 | 10
score on a scale
  Pre (T0) | 17.91 (3.33) | 17.10 (4.75)
  Mid-Treatment (T1): number analyzed (Participants) | 9 | 8
  Mid-Treatment (T1) | 14.11 (2.98) | 13.13 (4.82)
  Post (T2): number analyzed (Participants) | 7 | 8
  Post (T2) | 6.32 (4.24) | 7.38 (4.44)
  6 Month Fup (T4): number analyzed (Participants) | 6 | 6
  6 Month Fup (T4) | 4.67 (6.41) | 6.50 (4.59)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.62, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = 1.06, 95% CI 2-sided [-3.14 to 5.25]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.54, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 1.83, 95% CI 2-sided [-4.07 to 7.73]

6. Secondary Outcome: Mean Beck-Depression Inventory-II (BDI-II) Total Score in Modified Intent-to-Treat Patients and Partners
Description: The Beck Depression Inventory-II (BDI-II) is one of the most widely used self-report measures of depressive symptoms. It includes 21 self-report items. Total scores range from 0 to 63, and higher scores indicate higher levels of depressive symptoms
Time Frame: as for outcome 2
Population: Both patients and partners completed this measure. Participants who provided data were analyzed. Some participants provided partial data at study time points, explaining discrepancy(ies) between the mITT Participant Flow N and N analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 22 | 20
score on a scale
  Pre (T0) Patients: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients | 18.82 (8.53) | 19.50 (8.49)
  Mid-Treatment (T1) Patients: number analyzed (Participants) | 10 | 8
  Mid-Treatment (T1) Patients | 10.90 (6.79) | 14.88 (8.49)
  Post (T2) Patients: number analyzed (Participants) | 7 | 7
  Post (T2) Patients | 7.14 (4.22) | 12.00 (7.70)
  3 Month Fup (T3) Patients: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients | 7.33 (4.89) | 9.13 (7.53)
  6 Month Fup (T4) Patients: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients | 4.33 (4.27) | 7.43 (3.95)
  Pre (T0) Partners: number analyzed (Participants) | 11 | 10
  Pre (T0) Partners | 6.18 (4.75) | 6.00 (5.70)
  Mid-Treatment (T1) Partners: number analyzed (Participants) | 7 | 8
  Mid-Treatment (T1) Partners | 5.43 (5.03) | 5.75 (7.63)
  Post (T2) Partners: number analyzed (Participants) | 6 | 8
  Post (T2) Partners | 7.50 (8.04) | 5.88 (5.54)
  3 Month Fup (T3) Partners: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Partners | 8.00 (8.02) | 5.50 (6.50)
  6 Month Fup (T4) Partners: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Partners | 7.67 (9.65) | 5.29 (8.08)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.10, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = 4.80, 95% CI 2-sided [-0.91 to 10.51]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.76, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = 1.08, 95% CI 2-sided [-5.97 to 8.13]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.23, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 3.26, 95% CI 2-sided [-2.03 to 8.55]
Statistical Analysis 4: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.94, Mixed Models Analysis — Comparison of Partners at Post (T2); LS mean difference = -0.25, 95% CI 2-sided [-6.63 to 6.14]
Statistical Analysis 5: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.68, Mixed Models Analysis — Comparison of Partners at 3 Month Fup (T3); LS mean difference = -1.46, 95% CI 2-sided [-8.38 to 5.46]
Statistical Analysis 6: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.89, Mixed Models Analysis — Comparison of Partners at 6 Month Fup (T4); LS mean difference = -0.61, 95% CI 2-sided [-9.06 to 7.84]

7. Secondary Outcome: Mean Beck Anxiety Inventory-II (BAI-II) Total Score in Modified Intent-to-Treat Patients and Partners
Description: The Beck-Anxiety Inventory-II (BAI) is a self-report measure that assesses different aspects of the anxiety experience (e.g., physiological, cognitive, behavioral). The total score ranges from 0 to 63 with higher scores indicative of greater anxiety symptoms.
Time Frame: as for outcome 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 22 | 20
score on a scale
  Pre (T0) Patients: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients | 8.18 (4.92) | 13.40 (8.80)
  Mid-Treatment (T1) Patients: number analyzed (Participants) | 10 | 8
  Mid-Treatment (T1) Patients | 8.00 (5.46) | 12.25 (12.70)
  Post (T2) Patients: number analyzed (Participants) | 7 | 7
  Post (T2) Patients | 9.43 (7.02) | 5.71 (4.19)
  3 Month Fup (T3) Patients: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients | 5.33 (6.44) | 9.88 (9.30)
  6 Month Fup (T4) Patients: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients | 3.83 (4.12) | 4.71 (4.72)
  Pre (T0) Partners: number analyzed (Participants) | 11 | 10
  Pre (T0) Partners | 2.64 (3.44) | 6.00 (7.45)
  Mid-Treatment (T1) Partners: number analyzed (Participants) | 7 | 8
  Mid-Treatment (T1) Partners | 4.14 (5.76) | 9.75 (13.86)
  Post (T2) Partners: number analyzed (Participants) | 6 | 8
  Post (T2) Partners | 4.00 (3.29) | 6.13 (10.01)
  3 Month Fup (T3) Partners: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Partners | 2.50 (3.27) | 5.13 (8.48)
  6 Month Fup (T4) Partners: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Partners | 3.17 (4.17) | 2.14 (3.02)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.91, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = -0.41, 95% CI 2-sided [-7.61 to 6.79]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.20, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = 4.72, 95% CI 2-sided [-2.49 to 11.93]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.14, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 4.78, 95% CI 2-sided [-1.63 to 11.20]
Statistical Analysis 4: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.25, Mixed Models Analysis — Comparison of Partners at Post (T2); LS mean difference = 3.86, 95% CI 2-sided [-2.76 to 10.49]
Statistical Analysis 5: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.14, Mixed Models Analysis — Comparison of Partners at 3 Month Fup (T3); LS mean difference = 4.22, 95% CI 2-sided [-1.45 to 9.89]
Statistical Analysis 6: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.28, Mixed Models Analysis — Comparison of Partners at 6 Month Fup (T4); LS mean difference = 3.15, 95% CI 2-sided [-2.58 to 8.87]

8. Secondary Outcome: Mean Difficulties in Emotion Regulation Scale (DERS) Total Score in Modified Intent-to-Treat Patients and Partners
Description: The Difficulties in Emotion Regulation Scale is a 36-item self-report scale that assesses emotion regulation. Item responses range from 1 to 5, with a total score range of 36 to 180. Higher scores indicate more difficulties in emotion regulation.
Time Frame: as for outcome 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 22 | 20
score on a scale
  Pre (T0) Patients: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients | 85.73 (19.06) | 97.60 (25.36)
  Mid-Treatment (T1) Patients: number analyzed (Participants) | 10 | 8
  Mid-Treatment (T1) Patients | 77.60 (19.72) | 90.13 (23.34)
  Post (T2) Patients: number analyzed (Participants) | 7 | 7
  Post (T2) Patients | 79.00 (17.82) | 73.71 (16.68)
  3 Month Fup (T3) Patients: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients | 66.17 (21.25) | 74.88 (21.45)
  6 Month Fup (T4) Patients: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients | 66.00 (20.38) | 72.14 (18.46)
  Pre (T0) Partners: number analyzed (Participants) | 11 | 10
  Pre (T0) Partners | 76.18 (23.46) | 64.50 (16.22)
  Mid-Treatment (T1) Partners: number analyzed (Participants) | 7 | 8
  Mid-Treatment (T1) Partners | 65.86 (23.74) | 66.63 (17.48)
  Post (T2) Partners: number analyzed (Participants) | 6 | 8
  Post (T2) Partners | 69.67 (24.86) | 68.25 (19.65)
  3 Month Fup (T3) Partners: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Partners | 72.33 (24.47) | 66.00 (17.34)
  6 Month Fup (T4) Partners: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Partners | 69.17 (18.76) | 61.43 (16.40)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.85, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = 1.73, 95% CI 2-sided [-16.73 to 20.19]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.47, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = 7.94, 95% CI 2-sided [-13.59 to 29.48]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.37, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 9.79, 95% CI 2-sided [-11.50 to 31.08]
Statistical Analysis 4: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.97, Mixed Models Analysis — Comparison of Partners at Post (T2); LS mean difference = 0.36, 95% CI 2-sided [-19.31 to 20.03]
Statistical Analysis 5: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.52, Mixed Models Analysis — Comparison of Partners at 3 Month Fup (T3); LS mean difference = -5.88, 95% CI 2-sided [-23.85 to 12.09]
Statistical Analysis 6: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.68, Mixed Models Analysis — Comparison of Partners at 6 Month Fup (T4); LS mean difference = -3.55, 95% CI 2-sided [-20.33 to 13.23]

9. Secondary Outcome: Mean Partner Difficulties in Emotion Regulation Scale (DERS) Total Score in Modified Intent-to-Treat Patients and Partners
Description: The partner version of the Difficulties in Emotion Regulation Scale is an 8-item modified version of the DERS. It is a self-report scale that assesses perceptions of one's partner's emotion regulation ability and skills. Three items from the Impulse Control Difficulties (ICD) and 5 items from the Emotion Regulation Strategies (ERS) subscale were administered. Item responses range from 1 to 5 and the total score is the sum of the items. The total score range is 8 to 40. Higher scores indicate more (perceived) difficulties in one's partner's emotion regulation.
Time Frame: as for outcome 2
Population: Both patients and partners completed this measure. Participants who provided data were analyzed. Some participants provided partial data at study time points, further, one participant was no longer in a relationship for midpoint-6 month follow-up (T1-T4) assessments and thus, did not complete couple-based measures; this explains discrepancy(ies) between the mITT Participant Flow N and N analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 22 | 20
score on a scale
  Pre (T0) Patients: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients | 15.36 (5.52) | 16.60 (5.85)
  Mid-Treatment (T1) Patients: number analyzed (Participants) | 9 | 8
  Mid-Treatment (T1) Patients | 13.89 (5.58) | 19.38 (8.37)
  Post (T2) Patients: number analyzed (Participants) | 7 | 7
  Post (T2) Patients | 15.86 (4.14) | 16.71 (5.35)
  3 Month Fup (T3) Patients: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients | 13.83 (4.45) | 18.38 (6.99)
  6 Month Fup (T4) Patients: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients | 15.17 (6.91) | 18.29 (8.69)
  Pre (T0) Partners: number analyzed (Participants) | 11 | 10
  Pre (T0) Partners | 20.73 (8.60) | 15.40 (4.95)
  Mid-Treatment (T1) Partners: number analyzed (Participants) | 7 | 8
  Mid-Treatment (T1) Partners | 22.71 (10.40) | 16.63 (5.10)
  Post (T2) Partners: number analyzed (Participants) | 6 | 8
  Post (T2) Partners | 19.17 (8.84) | 15.75 (5.01)
  3 Month Fup (T3) Partners: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Partners | 21.17 (11.30) | 14.38 (4.60)
  6 Month Fup (T4) Partners: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Partners | 20.33 (9.67) | 12.71 (2.81)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.91, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = -0.27, 95% CI 2-sided [-5.02 to 4.47]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.07, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = 4.73, 95% CI 2-sided [-0.36 to 9.81]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.65, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 1.75, 95% CI 2-sided [-5.73 to 9.23]
Statistical Analysis 4: Comparison: CBT-E vs UNITE; Comparison of Partners at Post (T2); Test type: Superiority; p = 0.52, Mixed Models Analysis; LS mean difference = -2.05, 95% CI 2-sided [-8.21 to 4.12]
Statistical Analysis 5: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.07, Mixed Models Analysis — Comparison of Partners at 3 Month Fup (T3); LS mean difference = -6.62, 95% CI 2-sided [-13.74 to 0.51]
Statistical Analysis 6: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.03, Mixed Models Analysis — Comparison of Partners at 6 Month Fup (T4); LS mean difference = -6.64, 95% CI 2-sided [-12.73 to -0.56]

10. Secondary Outcome: Mean Dyadic Adjustment Scale (DAS-32) Total Score in Modified Intent-to-Treat Patients and Partners
Description: The Dyadic Adjustment Scale is a 32-item self-report scale that assesses the quality of the relationship as perceived by participants. The total score range is 0 to 151. Higher scores indicate higher dyadic adjustment within the relationship and greater relationship satisfaction.
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 22 | 20
score on a scale
  Pre (T0) Patients: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients | 112.27 (15.31) | 109.60 (18.84)
  Mid-Treatment (T1) Patients: number analyzed (Participants) | 9 | 8
  Mid-Treatment (T1) Patients | 115.44 (12.13) | 112.00 (18.50)
  Post (T2) Patients: number analyzed (Participants) | 7 | 7
  Post (T2) Patients | 117.29 (19.76) | 119.29 (14.04)
  3 Month Fup (T3) Patients: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients | 113.67 (23.96) | 112.75 (17.77)
  6 Month Fup (T4) Patients: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients | 114.17 (26.13) | 116.43 (15.98)
  Pre (T0) Partners: number analyzed (Participants) | 11 | 10
  Pre (T0) Partners | 110.27 (14.95) | 116.00 (16.75)
  Mid-Treatment (T1) Partners: number analyzed (Participants) | 7 | 7
  Mid-Treatment (T1) Partners | 112.14 (16.63) | 112.71 (14.31)
  Post (T2) Partners: number analyzed (Participants) | 6 | 7
  Post (T2) Partners | 111.17 (7.88) | 119.43 (16.00)
  3 Month Fup (T3) Partners: number analyzed (Participants) | 6 | 6
  3 Month Fup (T3) Partners | 110.67 (7.12) | 117.83 (17.93)
  6 Month Fup (T4) Partners: number analyzed (Participants) | 6 | 6
  6 Month Fup (T4) Partners | 112.50 (9.77) | 114.00 (21.36)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.90, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = 0.88, 95% CI 2-sided [-13.43 to 15.19]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.95, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = -0.64, 95% CI 2-sided [-18.95 to 17.66]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.89, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 1.37, 95% CI 2-sided [-17.17 to 19.90]
Statistical Analysis 4: Comparison: CBT-E vs UNITE; Comparison of Partners at Post (T2); Test type: Superiority; p = 0.39, Mixed Models Analysis; LS mean difference = 5.81, 95% CI 2-sided [-7.37 to 18.98]
Statistical Analysis 5: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.36, Mixed Models Analysis — Comparison of Partners at 3 Month Fup (T3); LS mean difference = 6.29, 95% CI 2-sided [-7.26 to 19.84]
Statistical Analysis 6: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.87, Mixed Models Analysis — Comparison of Partners at 6 Month Fup (T4); LS mean difference = -1.55, 95% CI 2-sided [-20.00 to 16.91]

11. Secondary Outcome: Mean Dyadic Adjustment Scale-Short Form (DAS-4) Total Score in Modified Intent-to-Treat Patients and Partners
Description: The Dyadic Adjustment Scale-Short Form (DAS-4) is a 4-item self-report scale that assesses the quality of the relationship as perceived by participants. The total score range is 0 to 21. Higher scores indicate higher dyadic adjustment within the relationship and greater relationship satisfaction.
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 22 | 20
score on a scale
  Pre (T0) Patients: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients | 15.91 (2.34) | 16.30 (2.87)
  Mid-Treatment (T1) Patients: number analyzed (Participants) | 9 | 8
  Mid-Treatment (T1) Patients | 17.33 (1.66) | 16.13 (2.70)
  Post (T2) Patients: number analyzed (Participants) | 7 | 7
  Post (T2) Patients | 16.71 (3.04) | 17.00 (2.83)
  3 Month Fup (T3) Patients: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients | 17.33 (2.42) | 16.13 (3.48)
  6 Month Fup (T4) Patients: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients | 17.00 (3.10) | 17.43 (2.76)
  Pre (T0) Partners: number analyzed (Participants) | 11 | 10
  Pre (T0) Partners | 15.82 (2.64) | 15.90 (3.11)
  Mid-Treatment (T1) Partners: number analyzed (Participants) | 7 | 8
  Mid-Treatment (T1) Partners | 15.86 (2.19) | 15.50 (1.93)
  Post (T2) Partners: number analyzed (Participants) | 6 | 8
  Post (T2) Partners | 16.67 (1.37) | 17.13 (2.17)
  3 Month Fup (T3) Partners: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Partners | 15.83 (2.23) | 17.25 (2.25)
  6 Month Fup (T4) Partners: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Partners | 16.00 (2.19) | 17.29 (2.14)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.84, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = 0.27, 95% CI 2-sided [-2.29 to 2.83]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.57, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = -0.82, 95% CI 2-sided [-3.66 to 2.01]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.67, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 0.6, 95% CI 2-sided [-2.15 to 3.35]
Statistical Analysis 4: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.63, Mixed Models Analysis — Comparison of Partners at Post (T2); LS mean difference = 0.46, 95% CI 2-sided [-1.43 to 2.35]
Statistical Analysis 5: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.21, Mixed Models Analysis — Comparison of Partners at 3 Month Fup (T3); LS mean difference = 1.44, 95% CI 2-sided [-0.82 to 3.70]
Statistical Analysis 6: Comparison: CBT-E; Test type: Superiority; p = 0.34, Mixed Models Analysis — Comparison of Partners at 6 Month Fup (T4); LS mean difference = 1.07, 95% CI 2-sided [-1.14 to 3.28]

12. Secondary Outcome: Mean Communication Patterns Questionnaire-Short Form (CPQ-SF) Subscale Scores in Modified Intent-to-Treat Patients and Partners
Description: The Communication Patterns Questionnaire-Short Form (modified for Binge-Eating Disorder) assesses how the couple communicates about binge-eating when the issue arises and when discussing the issue. Item responses range from 1 to 9. The three subscales measured are Self Demand/Partner Withdraw (3 items), Partner Demand/Self Withdraw (3 items), and Constructive Communication (3 items). The Demand/Withdraw subscales were combined and have a score range of 6 to 54 and the Constructive Communication subscale has a score range of 3 to 27. Higher (subscale) sum scores indicate more of those types of behaviors, respectively; high scores on the Demand/Withdraw and low scores on the Constructive Communication subscale are worse, respectively.
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 22 | 20
score on a scale
  Pre (T0) Patients, Demand/Withdraw subscale: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients, Demand/Withdraw subscale | 18.55 (6.65) | 20.70 (10.94)
  Mid-Treatment (T1) Patients, Demand/Withdraw subscale: number analyzed (Participants) | 9 | 8
  Mid-Treatment (T1) Patients, Demand/Withdraw subscale | 16.33 (8.90) | 18.38 (8.37)
  Post (T2) Patients, Demand/Withdraw subscale: number analyzed (Participants) | 7 | 7
  Post (T2) Patients, Demand/Withdraw subscale | 18.57 (9.62) | 15.29 (11.64)
  3 Month Fup (T3) Patients, Demand/Withdraw subscale: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients, Demand/Withdraw subscale | 12.50 (7.61) | 12.88 (6.83)
  6 Month Fup (T4) Patients, Demand/Withdraw subscale: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients, Demand/Withdraw subscale | 13.00 (5.93) | 13.43 (7.96)
  Pre (T0) Partners, Demand/Withdraw subscale: number analyzed (Participants) | 11 | 10
  Pre (T0) Partners, Demand/Withdraw subscale | 18.36 (8.09) | 14.50 (8.75)
  Mid-Treatment (T1) Partners, Demand/Withdraw subscale: number analyzed (Participants) | 7 | 8
  Mid-Treatment (T1) Partners, Demand/Withdraw subscale | 16.57 (8.32) | 16.50 (6.57)
  Post (T2) Partners, Demand/Withdraw subscale: number analyzed (Participants) | 6 | 8
  Post (T2) Partners, Demand/Withdraw subscale | 22.83 (9.79) | 12.25 (5.28)
  3 Month Fup (T3) Partners, Demand/Withdraw subscale: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Partners, Demand/Withdraw subscale | 14.00 (9.06) | 14.13 (6.85)
  6 Month Fup (T4) Partners, Demand/Withdraw subscale: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Partners, Demand/Withdraw subscale | 16.33 (6.28) | 14.71 (8.40)
  Pre (T0) Patients, Constructive Communication subscale: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients, Constructive Communication subscale | 18.45 (6.98) | 16.40 (4.67)
  Mid-Treatment (T1) Patients, Constructive Communication subscale: number analyzed (Participants) | 9 | 8
  Mid-Treatment (T1) Patients, Constructive Communication subscale | 17.56 (7.26) | 16.00 (5.24)
  Post (T2) Patients, Constructive Communication subscale: number analyzed (Participants) | 7 | 7
  Post (T2) Patients, Constructive Communication subscale | 19.86 (5.84) | 21.86 (4.22)
  3 Month Fup (T3) Patients, Constructive Communication subscale: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients, Constructive Communication subscale | 18.83 (9.33) | 20.38 (4.84)
  6 Month Fup (T4) Patients, Constructive Communication subscale: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients, Constructive Communication subscale | 18.33 (9.29) | 21.43 (3.64)
  Pre (T0) Partners, Constructive Communication subscale: number analyzed (Participants) | 11 | 10
  Pre (T0) Partners, Constructive Communication subscale | 15.18 (6.03) | 20.20 (3.97)
  Mid-Treatment (T1) Partners, Constructive Communication subscale: number analyzed (Participants) | 7 | 8
  Mid-Treatment (T1) Partners, Constructive Communication subscale | 19.57 (4.47) | 20.50 (3.46)
  Post (T2) Partners, Constructive Communication subscale: number analyzed (Participants) | 6 | 8
  Post (T2) Partners, Constructive Communication subscale | 20.83 (4.79) | 22.88 (2.95)
  3 Month Fup (T3) Partners, Constructive Communication subscale: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Partners, Constructive Communication subscale | 18.17 (6.40) | 20.75 (4.23)
  6 Month Fup (T4) Partners, Constructive Communication subscale: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Partners, Constructive Communication subscale | 20.33 (5.28) | 21.86 (4.41)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.50, Mixed Models Analysis — Demand/Withdraw score: Comparison of Patients at Post (T2); LS mean difference = -3.42, 95% CI 2-sided [-13.36 to 6.52]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.89, Mixed Models Analysis — Demand/Withdraw Score: Comparison of Patients at 3 Month Fup (T3); LS mean difference = -0.47, 95% CI 2-sided [-7.49 to 6.54]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.86, Mixed Models Analysis — Demand/Withdraw Score: Comparison of Patients at 6 Month Fup (T4); LS mean difference = -0.63, 95% CI 2-sided [-7.56 to 6.30]
Statistical Analysis 4: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.25, Mixed Models Analysis — Constructive Communication Score: Comparison of Patients at Post (T2); LS mean difference = 2.55, 95% CI 2-sided [-1.83 to 6.93]
Statistical Analysis 5: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.56, Mixed Models Analysis — Constructive Communication Score: Comparison of Patients at 3 Month Fup (T3); LS mean difference = 2.05, 95% CI 2-sided [-4.83 to 8.92]
Statistical Analysis 6: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.34, Mixed Models Analysis — Constructive Communication Score: Comparison of Patients at 6 Month Fup (T4); LS mean difference = 3.13, 95% CI 2-sided [-3.27 to 9.54]
Statistical Analysis 7: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.02, Mixed Models Analysis — Demand/Withdraw score: Comparison of Partners at Post (T2); LS mean difference = -10.24, 95% CI 2-sided [-19.05 to -1.42]
Statistical Analysis 8: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.98, Mixed Models Analysis — Demand/Withdraw score: Comparison of Partners at 3 Month Fup (T3); LS mean difference = -0.12, 95% CI 2-sided [-8.18 to 7.95]
Statistical Analysis 9: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.59, Mixed Models Analysis — Demand/Withdraw score: Comparison of Partners at 6 Month Fup (T4); LS mean difference = -2.20, 95% CI 2-sided [-10.10 to 5.70]
Statistical Analysis 10: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.16, Mixed Models Analysis — Constructive Communication Score: Comparison of Partners at Post (T2); LS mean difference = 2.41, 95% CI 2-sided [-0.99 to 5.82]
Statistical Analysis 11: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.12, Mixed Models Analysis — Constructive Communication Score: Comparison of Partners at 3 Month Fup (T3); LS mean difference = 3.94, 95% CI 2-sided [-1.05 to 8.93]
Statistical Analysis 12: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.34, Mixed Models Analysis — Constructive Communication Score: Comparison of Partners at 6 Month Fup (T4); LS mean difference = 2.26, 95% CI 2-sided [-2.35 to 6.87]

13. Secondary Outcome: Mean Eating Disorder Quality of Life Questionnaire (EDQOL) Total Score in Modified Intent-to-Treat Patients
Description: The Eating Disorder Quality of Life questionnaire is a self-report 25-item health-related quality of life questionnaire that measures the perceived extent to which the eating disorder affects the subject's quality of life in different domains. Item responses range from 0 to 4, with a possible score range of 0 to 100. Higher scores indicate lower quality of life.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 11 | 10
score on a scale
  Pre (T0) | 1.22 (0.58) | 1.38 (0.55)
  Mid-Treatment (T1): number analyzed (Participants) | 10 | 8
  Mid-Treatment (T1) | 0.86 (0.41) | 1.10 (0.44)
  Post (T2): number analyzed (Participants) | 7 | 7
  Post (T2) | 0.86 (0.45) | 0.73 (0.36)
  3 Month Fup (T3): number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) | 0.63 (0.51) | 0.52 (0.43)
  6 Month Fup (T4): number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) | 0.45 (0.65) | 0.51 (0.47)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.70, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = 0.09, 95% CI 2-sided [-0.35 to 0.53]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.90, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = -0.03, 95% CI 2-sided [-0.48 to 0.42]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.38, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = 0.25, 95% CI 2-sided [-0.31 to 0.82]

14. Secondary Outcome: Mean Problem-Solving/Communication Subscale Score of the Marital Satisfaction Inventory-Revised (MSI-R) in Modified Intent-to-Treat Patients and Partners
Description: This revised version of the Marital Satisfaction Inventory is a 150-item true/false self-report assessment of marital distress. For the purposes of this study, the investigators examined the Problem-Solving Communication scale (PSC - 19 items), which measures the inability to resolve differences in the relationship. PSC scores range from 0-19 with higher scores indicating poorer problem-solving communication skills.
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 22 | 20
score on a scale
  Pre (T0) Patients: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients | 5.64 (4.23) | 7.20 (5.65)
  Mid-Treatment (T1) Patients: number analyzed (Participants) | 9 | 8
  Mid-Treatment (T1) Patients | 6.22 (4.84) | 8.25 (5.01)
  Post (T2) Patients: number analyzed (Participants) | 7 | 7
  Post (T2) Patients | 6.14 (4.74) | 6.14 (5.64)
  3 Month Fup (T3) Patients: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients | 6.17 (4.45) | 7.00 (5.83)
  6 Month Fup (T4) Patients: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients | 6.17 (5.85) | 6.14 (3.85)
  Pre (T0) Partners: number analyzed (Participants) | 11 | 9
  Pre (T0) Partners | 9.18 (6.40) | 6.33 (5.72)
  Mid-Treatment (T1) Partners: number analyzed (Participants) | 7 | 8
  Mid-Treatment (T1) Partners | 7.14 (5.40) | 7.25 (6.61)
  Post (T2) Partners: number analyzed (Participants) | 6 | 8
  Post (T2) Partners | 8.50 (5.89) | 5.75 (5.55)
  3 Month Fup (T3) Partners: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Partners | 10.00 (5.62) | 6.00 (5.37)
  6 Month Fup (T4) Partners: number analyzed (Participants) | 6 | 6
  6 Month Fup (T4) Partners | 8.50 (5.21) | 4.00 (5.33)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.89, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = -0.33, 95% CI 2-sided [-5.10 to 4.43]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.85, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = 0.45, 95% CI 2-sided [-4.14 to 5.04]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.72, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = -0.85, 95% CI 2-sided [-5.54 to 3.85]
Statistical Analysis 4: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.29, Mixed Models Analysis — Comparison of Partners at Post (T2); LS mean difference = -3.05, 95% CI 2-sided [-8.73 to 2.63]
Statistical Analysis 5: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.08, Mixed Models Analysis — Comparison of Partners at 3 Month Fup (T3); LS mean difference = -4.69, 95% CI 2-sided [-9.90 to 0.51]
Statistical Analysis 6: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.19, Mixed Models Analysis — Comparison of Partners at 6 Month Fup (T4); LS mean difference = -3.29, 95% CI 2-sided [-8.23 to 1.65]

15. Secondary Outcome: Mean Affective Communication Subscale Score of the Marital Satisfaction Inventory-Revised (MSI-R) in Modified Intent-to-Treat Patients and Partners
Description: This revised version of the Marital Satisfaction Inventory is a 150-item true/false self-report assessment of marital distress. For the purposes of this study the investigators examined the 13-item Affective Communication scale (ACS), which assesses general communication. ACS scores range from 0-13 with higher scores indicating poorer affective communication skills.
Time Frame: as for outcome 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 22 | 20
score on a scale
  Pre (T0) Patients: number analyzed (Participants) | 11 | 10
  Pre (T0) Patients | 4.09 (3.36) | 4.30 (3.71)
  Mid-Treatment (T1) Patients: number analyzed (Participants) | 9 | 8
  Mid-Treatment (T1) Patients | 3.67 (3.84) | 5.13 (4.29)
  Post (T2) Patients: number analyzed (Participants) | 7 | 7
  Post (T2) Patients | 3.57 (4.39) | 2.57 (1.99)
  3 Month Fup (T3) Patients: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Patients | 4.17 (3.92) | 4.50 (3.34)
  6 Month Fup (T4) Patients: number analyzed (Participants) | 6 | 7
  6 Month Fup (T4) Patients | 4.33 (4.80) | 3.14 (2.48)
  Pre (T0) Partners: number analyzed (Participants) | 11 | 8
  Pre (T0) Partners | 4.36 (3.20) | 2.50 (2.14)
  Mid-Treatment (T1) Partners: number analyzed (Participants) | 7 | 7
  Mid-Treatment (T1) Partners | 4.00 (3.96) | 2.43 (2.37)
  Post (T2) Partners: number analyzed (Participants) | 6 | 8
  Post (T2) Partners | 3.83 (4.07) | 2.75 (3.20)
  3 Month Fup (T3) Partners: number analyzed (Participants) | 6 | 8
  3 Month Fup (T3) Partners | 3.83 (3.06) | 2.75 (2.60)
  6 Month Fup (T4) Partners: number analyzed (Participants) | 6 | 6
  6 Month Fup (T4) Partners | 4.00 (3.10) | 1.17 (1.33)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.41, Mixed Models Analysis — Comparison of Patients at Post (T2); LS mean difference = -1.20, 95% CI 2-sided [-4.08 to 1.67]
Statistical Analysis 2: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.84, Mixed Models Analysis — Comparison of Patients at 3 Month Fup (T3); LS mean difference = 0.33, 95% CI 2-sided [-2.87 to 3.54]
Statistical Analysis 3: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.50, Mixed Models Analysis — Comparison of Patients at 6 Month Fup (T4); LS mean difference = -1.21, 95% CI 2-sided [-4.76 to 2.34]
Statistical Analysis 4: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.52, Mixed Models Analysis — Comparison of Partners at Post (T2); LS mean difference = -1.09, 95% CI 2-sided [-4.43 to 2.24]
Statistical Analysis 5: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.30, Mixed Models Analysis — Comparison of Partners at 3 Month Fup (T3); LS mean difference = -1.38, 95% CI 2-sided [-3.96 to 1.21]
Statistical Analysis 6: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.03, Mixed Models Analysis — Comparison of Partners at 6 Month Fup (T4); LS mean difference = -2.52, 95% CI 2-sided [-4.78 to -0.25]

16. Secondary Outcome: Mean Client Satisfaction Questionnaire-8 (CSQ-8) Total Score in Modified Intent-to-Treat Patients and Partners
Description: Treatment acceptability was measured with the 8-item Client Satisfaction Questionnaire, a validated acceptability measure. Item responses run on a scale of 1 to 4, with a total score range of 8-32. Higher scores indicate greater treatment satisfaction (acceptability). An independent samples t test was conducted.
Time Frame: Post (after 16 weekly treatment sessions) (T2)
Population: Patients in CBT-E and UNITE, and partners in UNITE, completed this measure. CBT-E partners did not complete this measure as they did not receive any treatment. Participants who provided data were analyzed. Some participants provided partial data at study time points, explaining discrepancy(ies) between the mITT Participant Flow N and N analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT-E | UNITE
Number analyzed (Participants) | 7 | 15
score on a scale
  Post (T2) Patients: number analyzed (Participants) | 7 | 7
  Post (T2) Patients | 28.71 (3.64) | 29.24 (3.55)
  Post (T2) Partners: number analyzed (Participants) | 0 | 8
  Post (T2) Partners |  | 30.38 (2.56)
Statistical Analysis 1: Comparison: CBT-E vs UNITE; Test type: Superiority; p = 0.79, t-test, 2 sided — Comparison of Patients at Post (T2); Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-3.66 to 4.72]

17. Other Pre Specified Outcome: Couple Communication Measured by Observational Coding of Recorded Couple Conversations
Description: Couple communication will be assessed by rating of a 10-minute videotaped conversation in which the couple is asked to share thoughts, feelings, and concerns about some aspect of the patient's binge-eating disorder. Scoring will be based on the Couples Interaction Rating System (CIRS) and Social Support Interaction Rating System (SSIRS), observational coding systems that assess communication behaviors, affective expression, and supportive behavior.
Time Frame: From Pre-treatment through Follow-up
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Couple Interpersonal Problem-solving/Behavior Change Skills Measured by Observational Coding of a Recorded Couple Conversation
Description: Couple interpersonal problem-solving/behavior change skills will be assessed by rating of a 10-minute videotaped conversation in which the couple is asked to problem-solve on some aspect of the patient's binge-eating disorder and attempt to agree upon behavioral changes that they will make. Scoring will be based on the Couples Interaction Rating System (CIRS) and Social Support Interaction Rating System (SSIRS).
Time Frame: From Pre-treatment through Follow-up
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Partner-assisted Emotion Regulation Assessed With Vocally Encoded Emotional Arousal
Description: Two 10-minute video-taped interactions during which the couple is asked to share thoughts, feelings, and concerns about some aspect of the patient's binge-eating disorder and to problem-solve on some aspect of the patient's binge-eating disorder, respectively. Vocally encoded emotional arousal will be measured using fundamental frequency (f0) from patients' and partners' speech. F0 is a spectral analysis-based measure of speech prosody that refers to the lowest frequency harmonic of the speech sound wave, created by the opening and closing of the vocal folds while air flows outward from the lungs during speech production. Emotion regulation is indicated by one's ability to return to a stable set-point after being perturbed from that set-point. Stronger regulation is indicated by a faster return to the set-point. The range of fundamental frequency for speech in adult men and women is approximately 75-300hz.
Time Frame: From Pre-treatment through Follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the consent date to the 6-month follow-up.
Description: Adverse events (AEs) were collected by self-report, and participants, therapists, and staff shared any concerns. The investigators met biweekly with the Clinical Research Coordinator, and as needed, clinical supervisors or therapists to review participant safety. Any AE was required to be reported to the Data Safety and Monitoring Group (DSMG) immediately, and institutional review board (IRB), if appropriate. The DSMG met regularly to review safety data and maintained a record of AEs.
Groups:
- CBT-E Patients; CBT-E Partners: CBT-E is a trans-diagnostic cognitive behavioral individual therapy treatment for eating disorders. It has been shown to be effective in numerous controlled and open trials.
  CBT-E: CBT-E includes four stages: an introductory stage (psychoeducation, normalization of eating patterns, and symptom self-monitoring); a second, brief stage (review progress and formulate plans for the subsequent treatment phase); a third stage (elimination of dieting, reducing shape checking and avoidance behaviors, educating about mood tolerance, and targeting overevaluation of shape and weight); and the fourth stage (maintaining progress and minimizing relapse risk).
- UNITE Patients; UNITE Partners: UNITE is a manualized cognitive-behavioral couple therapy (CBCT) intervention that engages the couple to address the core psychopathology of BED.
  UNITE: UNITE includes three stages: early treatment (psychoeducation and understanding the couple's experience of BED within the relationship); mid-treatment (effective communication, interpersonal problem-solving, and emotion regulation skills), and late treatment (relapse prevention). Additional relevant topics may be covered including body image, weight stigma, weight and health concerns, and intimacy and sexuality issues.
Arm/Group | CBT-E Patients | CBT-E Partners | UNITE Patients | UNITE Partners
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Due to COVID-related issues, the recruitment target was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT03784820/Prot_SAP_001.pdf